CLINICAL TRIAL: NCT01105364
Title: Early Assessment of Anti-Angiogenic Treatment Efficacy in Advanced Renal Cancer by Using Contrast-Enhanced Sonography
Brief Title: Ultrasound in Assessing Antiangiogenic Treatment in Patients With Advanced Kidney Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, France (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: INCA-CIT07-FB-CREIN; CDR0000669914 (Registry Identifier: PDQ (Physician Data Query)); INCA-RECF0653-02; EUDRACT-2007-005627-15; PFIZER-INCA-CIT07-FB-CREIN
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2011-09

CONDITIONS: Kidney Cancer; Metastatic Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; liver metastases
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis; Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: antiangiogenesis therapy
Drug: stabilized sulphur hexafluoride microbubble-based contrast agent
Other: imaging biomarker analysis
Other: pharmacological study
Procedure: computed tomography
Procedure: magnetic resonance imaging

SUMMARY:
RATIONALE: Diagnostic procedures, such as contrast-enhanced ultrasound, may help measure a patient's response to treatment with drugs such as sunitinib malate, sorafenib tosylate, or bevacizumab, and allow doctors to plan better treatment.

PURPOSE: This clinical trial is studying ultrasonography in assessing antiangiogenic treatment in patients with advanced kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if contrast-enhanced ultrasonography (CEUS) study of target metastasis from renal cancer leads to early assessment of pharmacodynamic effects of antiangiogenic treatment in patients with advanced renal cancer.

Secondary

* To determine the association between functional changes of microvascularization and the target lesion by CEUS and the early objective response for this lesion indicated by the time to progression.
* To determine the association between functional changes of microvascularization and the target lesion by CEUS and the early objective response for this lesion indicated by the global survey.
* To determine the tolerance to antiangiogenic treatments in these patients.
* To determine the relationship between functional changes of microvascularization and the target lesion and the objective response for the other lesions (RECIST criteria) in cases of other metastasis other than the target lesion.

OUTLINE: Patients undergo contrast-enhanced ultrasonography (CEUS) before and after stabilized sulphur hexafluoride microbubble-based contrast agent injection. CEUS is done within 8 days prior to, 30 days after the first administration, and after 3 months of receiving antiangiogenesis treatment (e.g., sunitinib malate, sorafenib tosylate, or bevacizumab). Patients also undergo computed tomography and magnetic resonance imaging to evaluate tumoral targets.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced renal cancer
* Planning to receive antiangiogenic treatment
* Detection of a target hepatic metastasis that is visible, located, and sized with conventional sonography and CT scan and/or MRI

PATIENT CHARACTERISTICS:

* No active cardiac disease
* No severe arterial hypertension

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Lesion size (main diameter)
Arrival time within lesion
Time-to-peak
β parameter from enhancement curve
Density of microvessels at peak enhancement
Enhancement ratio between the lesion and the surrounding parenchyma at peak value
Determination of necrotic and viable volume
Tumoral response determined by RECIST criteria

SECONDARY OUTCOMES:
Time to progression
Global survey
Tolerance to antiangiogenic treatments
Objective response for non-target lesions

CONTACTS AND LOCATIONS:
Overall Officials: F. Bruyere, MD, Principal Investigator — Centre Hospitalier Universitaire Bretonneau de Tours
Locations (1):
- Centre Hospitalier Universitaire Bretonneau de Tours, Tours, France